CLINICAL TRIAL: NCT01766856
Title: Eustachian Tube Function as a Predictor of Myringoplasty/Tympanoplasty Outcome
Brief Title: Eustachian Tube Function and Myringoplasty/Tympanoplasty
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: University of Pittsburgh (Other)
Collaborators: Department of Pediatric Otolaryngology (Unknown)
Responsible Party: Principal Investigator, Margaretha L. Casselbrant, Professor of Otolaryngology, University of Pittsburgh
Other Study IDs: PRO12040564
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Tympanic Membrane Perforation
Keywords: perforation; tympanoplasty; myringoplasty; Eustachian tube function; tympanostomy tube
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children undergoing myringoplasty/tympanoplasty: child having repair of eardrum because of hole in eardrum after tube extruded or after tube removal
  Interventions: Other: Eustachian tube function testing

INTERVENTIONS:
Other: Eustachian tube function testing — Eustachian tube function testing will consist of some or all of the following tests: Inflation/Deflation test, Forced Response test, Compliance test,Valsalva, Toynbee and Sniffing

SUMMARY:
This study will determine whether the likely success of closing a hole in the eardrum can be predicted by testing Eustachian tube function. The Eustachian tube is a natural tube that connects the back of the nose with the middle ear. When a person goes up in an airplane and their ears "pop" or when one yawns and their ears "pop", that is the Eustachian tube opening. The Eustachian tube is responsible for keeping the air pressure in the middle ear the same as in the environment and keeping the middle ear free of fluid. It is thought that in children with middle-ear disease, the muscles that open the Eustachian tube do not work very well; this seems to get better in many children as they get older. It is thought that poor Eustachian tube function is the cause of failures when holes in the eardrum are patched and also for the recurrence of fluid in the middle-ear. The primary goal of this study is to see whether it can be predicted, based on testing Eustachian tube function before surgery, whether patching the eardrum will be successful and whether fluid will come back in the ear after it is patched.

DETAILED DESCRIPTION:
This study involves 1 visit to Children's Hospital of Pittsburgh of UPMC for Eustachian tube function testing and 2 visits, at approximately 6 months and at 12 months, after surgery to examine the ears.

Entry (Visit 1; approximately 40-60 minutes) At the entry visit, the child's medical history will be reviewed to ensure he/she is eligible for the study. The parent will be asked questions about their family, including family size, pets, medical history, tobacco smoke exposure, education and occupation, and living conditions. They will also be asked questions about their child, regarding such things as breastfeeding, daycare, tobacco smoke exposure and allergies, and a detailed history of middle-ear disease will be recorded. The child will have an examination of the ears, nose and throat.

Tympanometry will be done, which can help to tell whether there is fluid in the middle ear and whether there is an opening/hole in the eardrum. This is a common office procedure and is done by inserting a small probe (a rubber or plastic tube that measures ear pressure) half way into the ear canal and changing the pressure in the probe. That pressure change is small, can be felt but is rarely associated with any discomfort.

The function of the child's Eustachian tube on the side of the eardrum that is going to be patched will be tested. A small ear plug will be sealed partway into the child's ear canal. This plug is attached to a machine that can change the pressure in the ear and measure the pressure at which the Eustachian tube opens and closes, as well as the ease of airflow through the Eustachian tube and the ability to open the Eustachian tube during swallowing. The tests only require that the child not pull the ear plug from his/her ear and perform certain (age-appropriate) procedures designed to open his/her Eustachian tube such as swallowing with an open and pinched nose, blowing against a closed nose and deep breathing. The total time for testing is about 20 minutes and this period is broken into times of rest and times of tests. If the child has holes in both eardrums that are going to be repaired, testing may take 40 minutes.

After the entry testing: The child's ear surgeon will take a picture of the eardrum at the time of surgery to document the size of the hole. If the child does not require another surgical procedure after the surgery to close the eardrum because of failure of the hole to close or recurrence of ear problems such as infection or fluid in the ear, the child will have study visits for examination of the ears, nose and throat as well as tympanometry at approximately 6 months and 12 months after surgery. If he or she is being seen by the ear surgeon around these times, the study visit and their clinic visit can be done at the same time.

ELIGIBILITY:
Inclusion Criteria:

* 3-16 years old
* being scheduled for myringoplasty/tympanoplasty with removal of a patent tube or for repair of existing eardrum perforation remaining after a tube
* less than or equal to 8 weeks prior to surgery

Exclusion Criteria:

* syndromic or with craniofacial malformation (eg, Down syndrome, cleft palate)
* parent anticipates being unable to keep appointments (e.g., moving out of area)
* child unable to tolerate testing

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing myringoplasty/tympanoplasty for eardrum perforation after a tube or after a retained tube is removed.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Healing of perforation | 12 months
  Evidence of intact eardrum at 12 months after surgery
Recurrence of otitis media | by 12 months
  Recurrence of otitis media (acute otitis media and/or otitis media with effusion) by 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha L Casselbrant, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- ENT Research Center, Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No